CLINICAL TRIAL: NCT02975245
Title: Short Term Genetic Effects of Chemotherapy on Male Germ Cells
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kyle Orwig, Professor, University of Pittsburgh
Other Study IDs: STUDY20040140
Record Dates: First submitted 2016-11-21; First posted 2016-11-29 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cancer
Keywords: Male infertility; Germ cells; Chemotherapy; Sperm
MeSH Terms: conditions — Neoplasms; Infertility, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Semen sample
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (1):
- Men receiving chemotherapy: Semen collection and analysis
  Interventions: Procedure: Semen collection and analysis

INTERVENTIONS:
Procedure: Semen collection and analysis — Semen sample will be collected prior to the initiation of chemotherapy and one week after the first round of chemotherapy.

SUMMARY:
This study will determine the short-term effects of chemotherapy on sperm DNA.The study involves the collection of semen sample through ejaculation prior to initiation of chemotherapy and up to three time points after initiation of chemotherapy.

DETAILED DESCRIPTION:
While medical advances in the area of cancer treatment have successfully improved the overall detection and treatment of many cancers affecting men and women alike, these very treatment modalities can adversely affect their reproductive capacity.

Certain types of chemotherapy, such as alkylating agents, are notorious for placing patients at high risk for infertility. For men, the best recommendation for patients undergoing such therapy is to cryopreserve semen prior to initiation of chemotherapy. Unfortunately, this may not always occur. Some patients have been noted to present to discuss fertility preservation options after completing their first cycle of chemotherapy. In this situation, they will most likely still have sperm which was produced prior to chemotherapy that can be collected even if the stem cells producing the sperm have been damaged or destroyed. However, there are no national guidelines addressing this particular situation. Typically, physicians may advise men to avoid conception anywhere from three months to two years after the final dose of chemotherapy to ensure all exposed germ cells have passed through and only newly formed germ cells remain.

It is crucial to further assess the effects of chemotherapeutic agents on male germ cells in the short window of time between exposure and potential sterility. If a safe time frame could be determined to collect sperm after a single dose of chemotherapy, then these men could be given a second chance to retain their fertility potential.

ELIGIBILITY:
Inclusion Criteria:

* Be scheduled to undergo treatment with chemotherapeutic agents for a medical indication
* Be able to produce semen samples prior to chemotherapy and one week after first round of chemotherapy

Exclusion Criteria:

* Men who have previously been treated with chemotherapeutic agents.
* Men with significant oligospermia or azospermia.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Males between the ages of 18 and 50 who are scheduled to undergo chemotherapy for medical indication.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-02; Primary Completion 2025-04 (Actual); Study Completion 2025-04 (Actual)

PRIMARY OUTCOMES:
the differences in DNA between sperm collected before chemotherapy to sperm collected after the first round of chemotherapy using whole exome sequencing. | 5 years
  Sperm count test analyzes the health and viability of sperm, as it takes into account sperm number, motility, and morphology.

SECONDARY OUTCOMES:
changes in sperm quality from sperm collected before the initiation of chemotherapy to sperm collected after first round of chemotherapy using sperm count test. | 5 years
  Sperm count test analyzes the health and viability of sperm, as it takes into account sperm number, motility, and morphology.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Orwig, PhD, Principal Investigator — University of Pittsburgh/University of Pittsburgh Medical Center
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided